CLINICAL TRIAL: NCT03683381
Title: App-based Intervention for Treating Insomnia Among Patients With Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir H Pakpour, Supervisor, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR.QUMS.REC.1397.698
Record Dates: First submitted 2018-08-10; First posted 2018-09-25 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Epilepsy; Insomnia
MeSH Terms: conditions — Epilepsy; Sleep Initiation and Maintenance Disorders | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Patients in the intervention group will receive a 6-week app-based intervention to treat insomnia
  Interventions: Behavioral: Sleep Health
- patient education (Experimental): Participants in the patient education group will receive weekly information on insomnia symptoms
  Interventions: Other: Patient education

INTERVENTIONS:
Behavioral: Sleep Health — Participants in the intervention group will be provided with an application containing weekly instructions to improve sleep
  Arms: intervention
Other: Patient education — Participants in the Patient education group will receive weekly information on insomnia symptoms
  Arms: patient education

SUMMARY:
Sleep can affect frequency and occurrence of interictal spikes and occurrence, timing, and threshold of seizure. Epilepsy can worsen sleep architecture and severity of sleep disorders. Thus, a vicious cycle is set. Certain epilepsy syndromes are so intertwined with sleep that they are considered sleep-related epilepsies. Poor sleep in epilepsy is multifactorial and is worsened by poorly controlled seizures. App-delivered intervention has shown promise as a method to overcome health issues; however, the long-term effectiveness has not been proven in epileptic patients with chronic insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age
* diagnosis of epilepsy according to the International League Against Epilepsy criteria
* Self-report "moderate or severe" insomnia as indicated by a score of 15 or higher on the Insomnia Severity Index
* Can speak, understand, and write in Persian
* No surgery planned in the next 6 months
* Have access to an Android smartphone or a desktop computer with Internet access
* absence of major cognitive impairment or active psychiatric disorders

Exclusion Criteria:

* presence of a rapidly progressing neurological or medical disorder
* a diagnosis of mental retardation
* use of drugs or alcohol
* Untreated sleep apnea
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Insomnia symptoms | changes in ISI baseline , 1 month, 3 months and 6 months follow-up
  Isomnia symptom severity will be assessed using the Insomnia Severity Index
sleep hygiene behavior | changes in sleep hygiene behavior baseline , 1 month, 3 months and 6 months follow-up
  Sleep hygiene behaviour will use three items to measure how many days the participants had good sleep hygiene.
  behaviour.
objective sleep measure | changes in objective sleep baseline , 1 month and 6 months follow-up
  Sleep data is measured by Actigraphy (total minutes asleep, sleep effectiveness, sleep latency, awakenings). A wrist actigraph will be worn by the patients for 7 consecutive days.

SECONDARY OUTCOMES:
Psychological predictors of sleep hygiene behavior (attitude, habit, self monitoring, self control, perceived behavior control | changes from baseline , changes from baseline , 1 month and 6 Months follow-up
  psychological predictors of sleep hygiene behavior will be assessed using a using a self-reported measure. All items are rated on a Likert-type scale, ranging from 1 to 5.
Health related Quality of life | changes from baseline, changes from baseline , 1 month and 6 Months follow-up
  quality of Life in Epilepsy (QOLIE-31) will be used to assess quality of life
Anxiety and Depression | changes from baseline , changes from baseline , 1 month and 6 Months follow-up
  Zigmond and Snaith developed the 14-item HADS to measure the anxiety (7 items) and depression (7 items) of patients with both somatic and mental problems. The response descriptors of all items are Yes, definitely (score 3); Yes, sometimes (score 2); No, not much (score 1); No, not at all (score 0); except for items 7 and 10, which are scored reversely. A higher score represents higher levels of anxiety and depression: a domain score of 11 or greater indicates anxiety or depression; 8-10 indicates borderline case; 7 or lower indicates no signs of anxiety or depression. The two-factor framework of the HADS has been supported in epileptic patients.

CONTACTS AND LOCATIONS:
Locations (4):
- Iran (4):
  - Booali Sina Hospital, Qazvin
  - Shahid Rajaie Hospital, Qazvin
  - Firoozgar Hospital, Tehran
  - Mollasadra Neurology Clinic, Tehran

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Ahorsu DK, Lin CY, Imani V, Carlbring P, Nygardh A, Brostrom A, Hamilton K, Pakpour AH. Testing an app-based intervention to improve insomnia in patients with epilepsy: A randomized controlled trial. Epilepsy Behav. 2020 Nov;112:107371. doi: 10.1016/j.yebeh.2020.107371. Epub 2020 Aug 27. PMID 32861897